CLINICAL TRIAL: NCT02580643
Title: Prospective Post-Market Data Collection on Patients With Knee Osteoarthritis and Treated With nSTRIDE Autologous Protein Solution (REGP-22-00)
Brief Title: Prospective Post-Market Data Collection on Patients With Knee OA and Treated With nSTRIDE APS
Acronym: PROGRESS III
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: BBIO.CRNSAPS002.15
Record Dates: First submitted 2015-10-19; First posted 2015-10-20 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Autologous Protein Solution; Osteoarthritis; Intra-articular Injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- APS Injection: Autologous Protein Solution
  Interventions: Biological: APS

INTERVENTIONS:
Biological: APS — intra-articular injection

SUMMARY:
This study will document treatment effects, changes in quality of life, procedure complications, adverse events, healthcare resource utilization, and further needed intervention(s) following treatment with nSTRIDE autologous protein solution. This study will also allow for the documentation of the same parameters following multiple injections of autologous protein solution to treat knee osteoarthritis.

DETAILED DESCRIPTION:
Clinical trials have, in general, formally demonstrated the effectiveness and safety of various autologous therapies for the treatment of knee OA. Differences in the processing of autologous therapies can yield substantial differences in the resulting output. It appears that the safety of autologous therapies is roughly equivalent across different processing methods. However, making generalizations regarding the effectiveness across these autologous therapies is more complicated. Thus, each autologous therapy requires independent efficacy evaluation. nSTRIDE APS has been shown to decrease pain, increase function and have a favorable safety profile in a small pilot trial. However, demonstration of the treatment effects in a more heterogeneous population is lacking. Further, neither the effect time course nor the utility of multiple injections has been documented. This study will allow for low burden, efficient data collection in a larger heterogeneous population of persons suffering from knee OA. The study will document the treatment effects and timeline of treatment effects for nSTRIDE APS following single or repeated injections.

ELIGIBILITY:
Inclusion Criteria:

* OA of one or both knees as diagnosed by the treating physician
* At least 18 years of age
* Willing and able to comply with the study procedures
* Signed informed consent form

Exclusion Criteria:

* Any systemic inflammatory condition ( e.g., rheumatoid arthritis)
* Active malignancy at time of injection
* Pregnant at time of injection
* Lactating at the time of injection
* Knee joint infections or skin diseases or infections in the area of the injection site.
* Leukemia, metastatic malignant cells, or who are receiving chemotherapeutic treatment
* Participating in another device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with bilateral or unilateral knee OA will be prospectively enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Knee pain and function | Through 12 months
  Quantify and characterize the percentage of OMERACT-OARSI high improvement in pain responders at all post-injection time points. OMERACT-OARSI high improvement in pain responders are defined as subjects who show a 50% improvement in the KOOS pain sub-scale score and an absolute improvement of at least 20 points on the KOOS pain subscale score.

SECONDARY OUTCOMES:
Characterize the time from the initial nSTRIDE injection to subsequent nSTRIDE injection(s) or other intrusive treatment. | Through 12 months
Numeric Rating Scales (NRS) | Evaluated at 2 and 4 weeks and 3, 6 and 12 months
  Quantify the change in knee pain, stiffness and function
European Quality of Life 5 Dimensions 3 Levels (EQ-5D-3L) | Evaluated at 2 and 4 weeks and 3, 6 and 12 months
  Quantify the change in quality of life
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Evaluated at 2 and 4 weeks and 3, 6 and 12 months
  Quantify changes in pain, symptoms, activities of daily life, engagement in sports and recreation and quality of living
Procedural complications and adverse events | Through 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- BMI Bishops Wood Hospital, Northwood, United Kingdom